CLINICAL TRIAL: NCT03108612
Title: Exactitud diagnóstica Del Instrumento Análisis de Carga de Trabajo Para Identificar Riesgos Laborales en Trabajadores Con Trastornos músculo esqueléticos de Extremidades Superiores Que se evalúan en la Asociación Chilena de Seguridad.
Brief Title: Diagnostic Value of Workload Analysis Instrument to Detect Occupational Risks of Upper Limb Musculoskeletal Conditions
Acronym: ACT-ACHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medwave Estudios Limitada (Other)
Collaborators: Asociación Chilena de Seguridad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 203-2016
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2017-12

CONDITIONS: Musculoskeletal Disease; Occupational Exposure
Keywords: diagnostic accuracy; upper limb
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Participants are enrolled consecutively in the occupational health care clinic. After signing the informed consent form, the evaluators administer the index diagnostic test (WAI). Subsequently, the study participants are referred to the gold standard (EPT). Study participants, WAI evaluators and EPT evaluators are blinded to the results of the other test.
Masking Description: The care providers that administer the index test and the EPT assessment are not masked. However, the outcomes assesors of the EPT (gold standard) are masked to the results of the WAI (index test). The adminstrators of the WAI are unaware of the EPT result, as this evaluation is conducted after the application of the index test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Intervention: Análisis de carga de trabajo (ACT)
  Interventions: Diagnostic Test: Análisis de carga de trabajo (ACT)

INTERVENTIONS:
Diagnostic Test: Análisis de carga de trabajo (ACT) — Semi-structured interview for detecting possible occupational etiology of an upper limb musculoskeletal disease that has been reported (by the worker) as possibly of occupational origin. The instrument is called Workload Analysis Instrument (WAI) or Análisis de Carga de Trabajo (ACT).
  Other Names: Workload Analysis Instrument (WAI)

SUMMARY:
The aim of the study is to evaluate the diagnostic accuracy of an instrument (semi-structured interview) called Workload Analysis Instrument (WAI) (Análisis de Carga de Trabajo ACT), in detecting the presence of occupational risk in patients presenting an upper-limb musculoskeletal disorder. The test instrument was developed by Asociación Chilena de Seguridad (ACHS). This instrument will be applied to the worker when he or she visits the ACHS health care facility. The test administration is performed by an ergonomics specialist previously trained in WAI. WAI is the index test and the gold standard will be the Estudio de Puesto de Trabajo (EPT) resolution. The hypothesis of the study is that WAI is able to correctly label the occupational origin (rule in or rule out) of an upper-limb musculoskeletal disorder. Sensitivity, specificity and positive predictive value will be established.

DETAILED DESCRIPTION:
This is a cross sectional and prospective study where both the application of the index and reference instruments will be performed after the complete planning of the study.

Sample size was calculated assuming 90% sensitivity and 80% specificity of the WAI, based on experience with a similar instrument prior to WAI and on which WAI is built, which was used at the Hospital del Trabajador. For an absolute precision of 5%, the necessary sample size of people who actually have a work-related illness and those who do not actually have that origin should be 246. If 6% preciiosion is accepted that sample size should be 171.

Prevalence of ULMD qualified as from occupational origin is under 10% among patients who consult at the centers of the Metropolitan Region, according to the ACHS. Thus, the calculated final sample was approximately 1700 patients.

According to the project's budget, 900 applications of the WAI are to be planned.

The study will successively recruit patients: up to 246 true positives or 900 patients (whichever is reached first).

It is estimated that 75 WAI evaluations could be performed per month, with an average of 3.4 per day. Consequently, the sample of 900 would be achieved after 12 months.

FLOW OF PATIENTS Patients will be recruited in an ad hoc facility at the Hospital del Trabajador located in the Metropolitan Region.

Entry of a participant:

Each worker / patient who consults the facility or an emergency center of the ACHS agencies with a claim of professional illness involving a musculoskeletal disorder of the upper extremity (ULMD), within a pre-established range of time in a day and on pre-established days of the week, will be recruited for the study. The worker must voluntarily file a claim.

Derivation All consecutive workers with a suspicion of ULMD should be referred to the study. Once the attending physician verifies the patient meets the inclusion criteria, he or she will immediately refer the patient to the WAI evaluation without previously providing any information about the purpose of the study.

If for work reasons or force majeure the worker cannot immediately go to the place where the WAI evaluator is, an appointment will be made for another day according to the worker's availability. The rest of the medical treatment and other referrals will be indicated according to the regular medical procedure, thus preventing this new evaluation (WAI) from interfering with the patient's usual treatment.

Informed consent process:

Informed consent will be asked by the same evaluator. The process will be carried out in a room designated by the ACHS protecting the privacy of the participant. In this contact, the evaluator will spend approximately 10 minutes explaining the study objectives and asking for consent. Afterwards, the patient must read the informed consent document and he may refuse, doubt or accept to participate. In case of doubt the evaluator will inform the patient that one of the researchers will contact him or her within the next 24 hours and, if necessary, another appointment will be scheduled.

If the patient accepts immediately, he or she must sign the informed consent form and the evaluator will then proceed to the application of the WAI.

Evaluators:

For this study external personnel to the ACHS (evaluators) will be contracted and supervised by Medwave Estudios Limitada, and trained by the ACHS. Hired evaluators must be titled Kinesiologists with postgraduate experience in Ergonomics or Occupational Health.

Application of the instrument:

The WAI will be applied in the office designated by the ACHS. The evaluator will have approximately 30-45 minutes for this interview, in which he must collect all the necessary information. Application of the instrument will be done in accordance with the WAI manual prepared by the ACHS Workforce Survey team of evaluators.

Equipment and materials The room where the WAI is applied must be provided with a table and at least one chair with enough comfort for the patient to be seated during the duration of the interview and for the interviewer to ask the questions, listen to the answers and translate them into the document form which must be available in digital format.

MEASUREMENTS The general background of the worker and his place of work will be evaluated, as well as the worker´s sociodemographic characteristics. For the description of his work the occupational history and the type of work that he carries out will be evaluated emphasizing about schedules and rest arrangements. Job description will emerge from the detailed interview, considering tasks and times of effective and total work, breaks and overtime. The evaluator must not make a diagnostic hypothesis about the occupational origin of the illness.

WAI INTERPRETATION Once the WAI evaluation is obtained, it should be sent in the pre-established digital format to the ACHS office where it will be reviewed by a professional evaluator from the ACHS staff who must not be part of the final Qualification committee.

It is very important for a diagnostic accuracy study to preserve the masking of people who apply or interpret the instruments of the study in each stage of its conduction. The ACHS will have special responsibility in helping to maintain the masking.

The final professional evaluator (ACHS) must issue an opinion with three possibilities: 1) possible occupational origin, 2) discarded occupational origin and 3) doubtful. This final result of the WAI must be available not later than 15 business days, always before the result of the final evaluation (gold standard). Once the opinion is issued, each WAI will be sent to the Medwave Estudios Limitada headquarters for data processing and analysis.

TRAINING Training on the use of the WAI will be carried out by ACHS staff, led by the kinesiologist Patricia Ferreira. They were in charge of the preparation of the WAI and its manual. This training will take place during the month of April.

PILOT Once the approval of the Ethics Committee is obtained, and the WAI evaluators trained, we will proceed to perform the pilot phase whose objective will be to gauge all the inconveniences that emerge during the application of the instrument. The pilot will be carried out in the same facilities prepared for the study. Patients will meet the same inclusion criteria as those to be used in the study.

ABOUT THE GOLD STANDARD (WORKPLACE STUDY AND QUALIFICATION COMMITTEE) Patients who arrive for consultation with ACHS physicians for ULMD with a claim of work origin must undergo a "qualification process that includes several activities that the governing bodies must fulfill in order to determine the occupational or common origin of the diseases allegedly of professional origin" as set out in Circular 3241 of the Superintendence of Social Security, Chile, dated July 27, 2016. This circular:" instructs the administering agencies of Law Insurance 16744 on the protocol of minimum standards of evaluation that must be complied in the process of qualifying the origin of the diseases denounced as professionals ".

The qualification process will begin with the presentation of an individual claim of Professional Illness by the employer, the worker, their beneficiaries or others consigned in the circular. It includes a specific study of the workplace and must end with the final result given by a Qualification Committee which must determine the common or labor origin of the condition.

All evaluations must be carried out by professionals with specific competencies. - The study of workplace consists of the detailed analysis by observation in the field, the characteristics and environmental conditions in which a particular worker performs his job and the activities, tasks or operations that he performs. The qualification process must be concluded in full within a maximum period of 30 calendar days from the submission of the Individual Claim for Occupational Disease.

All of the above means that for each subject evaluated by the WAI, the final opinion of the Qualification Committee would have a maximum of 30 days.

The opinion of the Qualification Committee is the gold standard of the study for the definition of whether or not it is a pathology of possible occupational origin.

Once obtained the opinion of the Qualification Committee, the counterpart of the ACHS, coordinated in this case by Patricia Ferreira, will be in charge of weekly reports to the central office of data analysis located in Medwave Estudios. In this office, the data will be received by Matías Goyenechea, or whom he appoints. If, after a week has elapsed, no information has been received, the reception manager will monitor what happened during that time.

Data processing includes a database with all relevant data obtained from the WAI and the final result. Statistical analysis comprises the estimation of sensitivity, specificity and predictive values with their corresponding confidence intervals. Estimations will be made for the final diagnosis (occupational origin or not) as a whole and for each of the upper limbs segments considered where possible.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 and in a company affiliated to Asociación Chilena de Seguridad
* Suspicion of occupational origin of upper limb musculoskeletal disorder and have a registered claim of occupational origin of reported disorder (DIEP form)
* Disorder must be included in the following CIE-10 list: Trigger Finger ICD-10 code: M65.3; Flexor and extensor wrist tendinitis ICD-10 code: M65.8; Radial styloid tenosynovitis [de Quervain] ICD-10 ICD-10 code: M65.4; Carpal Tunnel Syndrome ICD-10 code: G56.0; Elbow Epitrocleitis ICD-10 code: M77.0; Epicondylitis ICD-10 code: M77.1; Shoulder tendinopathy of rotator cuff ICD-10 code: M75.1; Tendinitis bicipital ICD-10 code: M75.2; Subacromial bursitis ICD-10 code: M75.5

Exclusion Criteria:

* Not consulting within the study recruitment timetable for a consecutive sample
* Patients with physical limitations that preclude administering the instrument
* Patients with prior diagnosis of the included disorder (see above)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Occupational origin of upper limb musculoskeletal disorders | Participants are only assessed once when they are interviewed with the WAI. Final outcomes are obtained without the participant.
  Each patient´s disorder is classified as positive (occupational origin) or negative (non-occupational origin) by the index instrument and then by the gold standard. There are four possible main outcomes: true positive, true negative, false positive, false negative. Both the index instrument and the gold standard may yield a doubtful result.

CONTACTS AND LOCATIONS:
Overall Officials: Vivienne C. Bachelet, MD, MSc, Study Chair — Medwave Estudios Limitada
Locations (1):
- Hospital del Trabajador de la Asociación Chilena de Seguridad, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
The IPD will be anonymized in an Excel database. Permission to share with other investigators will be requested to the overseeing regulatory authority (Superintendencia de Seguridad Social). At the present time we cannot commit to sharing data without governmental approval.